CLINICAL TRIAL: NCT02878460
Title: ORI2 : ORI for hyperOxia Reduction in ICU
Acronym: ORI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-P2016-04; 2016-A01026-45 (Registry Identifier: ID RCB ANSM)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Intensive Care Units
Keywords: HYPEROXIA; MECHANICAL VENTILATION; OXYGEN RESERVE INDEX
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen Saturation; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monitoring with ORI + SpO2 (Experimental): Patients receive the regular monitoring with SpO2, but in this group, the ORI parameters is shown on the scope.
  Lower and upper SpO2 limits are prescribed for each patient.
  Interventions: Other: monitoring with ORI + SpO2
- monitoring with SpO2 (Other): Patients receive the regular monitoring; the ORI parameters is not shown (but it is recorded each time a blood gas is drown).
  Lower and upper SpO2 limits are prescribed for each patient.
  Interventions: Other: monitoring with SpO2

INTERVENTIONS:
Other: monitoring with ORI + SpO2 — If ORI is equal to 0.00, the FiO2 (or oxygen flow) is not changed. if ORI is ≥ 0.01, Nurses must decrease the FiO2 (or oxygen flow) by 10%, until ORI is =0.
  if SpO2 is < lower individualized limit, FiO2 (or oxygen flow) is increased by 10%, if it happens twice, doctors are called.
  Other Names: ORI group
  Arms: monitoring with ORI + SpO2
Other: monitoring with SpO2 — If SpO2 is below the upper individualized limit, the FiO2 (or oxygen flow) is not changed.
  If SpO2 is equal or above this limit, Nurses must reduce the FiO2 (or oxygen flow) by 10% every 10 minutes until SpO2 is ≤ upper individualized limit, with FiO2≥25 %.
  if SpO2 is < lower individualized limit, FiO2 (or oxygen flow) is increased by 10%, if it happens twice, doctors are called.
  Other Names: Control group
  Arms: monitoring with SpO2

SUMMARY:
Recently, hyperoxia has been recognized as being potentially deleterious for critically ill patients, with increased duration of mechanical ventilation and even with increased mortality rates. This could be related to pulmonary lesions (including notably atelectasis) but also to increased tissue damage and organ dysfunctions, secondary to increased/induced oxidative stress. At last higher FiO2 led to "over-consumption" of oxygen and therefore to additional costs. Usually, FiO2 and oxygen flows are modified according to the monitoring of SpO2. But, it has also been recognized that modifying FiO2 (and oxygen flows) according to SpO2 monitoring is not routinely (or easily) done. Indeed, nurses (and doctors) are reluctant to reduce oxygen flows when everything appear under control.

The ORI (Oxygen Reserve Index) is an index measured using non-invasive SpO2 sensors (Rainbow sensors- MASIMO) that evaluates non-invasively PaO2 (partial pressure of oxygen). An ORI ≤0 indicates that PaO2 is less than 100 mmHg. When ORI increases (i.e. ORI≥0.01) PaO2 is higher than 100 mmHg. This index increases up to 1. ORI between 0.01 and 1 indicates that PaO2 is probably between 100 and 200 mmHg. Thus, monitoring critically ill patients using the ORI, may help identifying when PaO2 is high and when FiO2 (or oxygen flows in non-intubated patients) may be reduced. This could help reducing the time with hyperoxia (i.e. PaO2 ≥100 mmHg or ≥80 mmHg).

The purpose of this feasibility study is to evaluate if the use of ORI can help to decrease length of moderate hyperoxia (PaO2>100mmHg) in critically ill patients, in comparison with monitoring the SpO2 only.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in ICU of Angers hospital
* Patient intubated and mechanically ventilated for an expected period of at least 2 days

Inclusion is to achieve within 6 hours after admission (for admitted patients intubated ) or at the time of intubation (for non- intubated patients on admission )

Exclusion Criteria:

* Pregnant Woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Percentage of days with moderate hyperoxia | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The primary endpoint is the percentage of days with moderate hyperoxia. Moderate hyperoxia is defined by a PaO2> 100 mmHg - measured on blood gases obtained in usual practicePaO2 will be followed by the inclusion until the end of mechanical ventilation or D28 or ICU discharge. The percentage of days with moderate hyperoxia is (number of days of moderate hyperoxia / number of days of oxygen therapy) x100. The follow up will occurs from inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge

SECONDARY OUTCOMES:
Minimum and maximum daily FiO2 | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoints are the minimum and maximum daily FiO2, obtained by respirator in each group. FiO2 will be followed by the inclusion until the end of oxygenotherapy or D28.
Minimum and maximum daily PaO2 | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoints are the minimum and maximum daily PaO2, (measured by blood gases obtained in usual practice ) . PaO2 will be followed by the inclusion until the end of oxygenotherapy or D28.
Length of mechanical ventilation | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoint is the length of mechanical ventilation, (unit: day number)
Number of day with PaO2 equal or above to 80 mmHg | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoint is the number of the day where patient is mechanically ventilated and has a PaO2 equal or above to 100 mmHg and 80 mmHg . PaO2 is measured by blood gases obtained in usual practice . this outcome will be followed by the inclusion until the end of mechanical ventilation or D28.
Number of hypoxemia episode | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoint is the number (in day) of hypoxemia (defined by PaO2<60 mmHg - measured by blood gases obtained in usual practice). PaO2 will be followed by the inclusion until the end of oxygenotherapy or D28.
Number of day without mechanical ventilation at D28 | inclusion to D28
  The secondary endpoint is the number of day without mechanical ventilation at D28. It will be followed by the inclusion until D28.
Number of atelectasis episodes requiring specific medical care (that means fibro-aspiration or posture of patient) | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoint is the number of atelectasis episodes requiring specific medical care. It will be followed by the inclusion until the end of mechanical ventilation or D28.
Average daily PaO2 | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The primary endpoint is the average daily PaO 2 in each group (measured by blood gases obtained in usual practice ) . PaO2 will be followed by the inclusion until the end of oxygenotherapy or D28.
Number of moderate hypoxemia hours | inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  this outcomes follows the formula: Moderate hypoxia (in hours) = a + b. With a = the sum of the durations (in hours) between two GDS having a PaO2> 100mmHg and b = the sum of the half times (in hours) between a GDS having a PaO2> 100mmHg and a GDS having a PaO2 ≤ 100mmHg
Maximum ORI values during pre-oxygenation before a endotracheal aspiration | At each pre-oxugenation before a endotracheal aspiration occurs from inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The secondary endpoint is the maximum ORI values during pre-oxygenation before a endotracheal aspiration
Minimum SpO2 within 15 minutes following a endotracheal aspiration | At each endotracheal aspiration occurs from inclusion to the end of mechanical ventilation or Day 28 if patient is still mechanically ventilated or ICU discharge
  The primary endpoint is the minimum SpO2 within 15 minutes following a endotracheal aspiration, with or without recruitment maneuver.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lasocki S, Brochant A, Leger M, Gaillard T, Lemarie P, Gergaud S, Dupre P. ORI monitoring allows a reduction of time with hyperoxia in critically ill patients: the randomized control ORI2 study. Intensive Care Med. 2019 Nov;45(11):1661-1662. doi: 10.1007/s00134-019-05732-9. Epub 2019 Aug 13. No abstract available. PMID 31410497